CLINICAL TRIAL: NCT03614208
Title: Effects of an Individualized, Home-based Exercise Program for the Patient With Systemic Sclerosis, on Exercise Capacity, Hand Mobility and Quality of Life: a Randomized, Controlled Study.
Brief Title: Individualized Home-based Exercise Program for Patient With Systemic Sclerosis.
Acronym: ESSE2016
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Marcello Ferrari, Professor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESSE2016
Record Dates: First submitted 2018-07-26; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Systemic Sclerosis
Keywords: Systemic sclerosis; Home based rehabilitation; Quality of life; Hand mobility; Exercise capacity
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: Single blind RCT with two parallel group
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-care rehabilitation group (HCRG) (Experimental): The home-based exercise program consists of aerobic exercise on a stationary bike, muscular endurance training of the upper limb and stretching exercises for finger joint motion. The exercise on the stationary bike and muscular endurance training will be performed on alternate days, three times a week. For finger stretching the patients will be directed to perform it every day, both in the morning and in the evening.
  During the rehabilitation period, the patients will report each day on a diary for each type of exercise. They received a phone call monthly, only for the first 3 months, to encourage them about the adherence and investigate any problems with the exercise program.
  Interventions: Behavioral: Home-care rehabilitation group (HCRG)
- Control group (No Intervention): Control group was encouraged to perform the generic aerobic physical activity at the baseline. Also, they received a monthly phone call, only for the first 3 months, to encourage them about the importance of doing aerobic exercise.

INTERVENTIONS:
Behavioral: Home-care rehabilitation group (HCRG) — The exercise program consists of aerobic exercise on a stationary bike, muscular endurance training of the upper limb and stretching exercises for finger joint motion. The exercise on the stationary bike and muscular endurance training will be performed on alternate days, three times a week.
  Other Names: Experimental group
  Arms: Home-care rehabilitation group (HCRG)

SUMMARY:
Systemic sclerosis (SSc) is an uncommon chronic rheumatic disease with an unknown cause and unpredictable course. The inability, in addition to easy fatigability, starts a vicious circle that leads to a fast deterioration of physical conditions that cause a reduction of aerobic exercise capacity and, consequently, of health-related quality of life (HRQoL). Aerobic exercise has already been shown to be safe and effective in improving exercise capacity and HRQoL of patients with chronic cardiovascular and pulmonary diseases. However, few studies have evaluated the role of specific exercise programs on the muscular impairment in SSc. Nevertheless, the results obtained in preliminary reports are promising, and, for these reasons, the management of muscular impairment in SSc could include an appropriate rehabilitation program besides pharmaceutical and surgical treatments.

The primary aim of this study will be to evaluate the effect of an individualized exercise program performed at home on aerobic capacity evaluated by 6 minutes walking test.

Secondary aims will be to evaluate: 1- VO2max, measured by cardiopulmonary test; 2- the effect of the same program on the muscular strength of upper and lower limbs; 3- the efficacy of a self-administered stretching program for finger joint motion. Secondary aims will be also 1-to ascertain whether a comprehensive exercise program may affect, besides physical function, HRQoL; 2- and to evaluate the adherence during two periods of three months, one whit and one without supervision and reinforcement by a phone call.

All the patients with a diagnosis of SSc, according to the criteria of American College of Rheumatology (ACR), who attended the Rheumatologic outpatient clinic of our institution will be evaluated in order to participate in the rehabilitation program. The pneumological examination and two days of screening and testing will take place at the outpatient's clinic of Respiratory Medicine and Sport of our institution.

DETAILED DESCRIPTION:
This will be a randomized, controlled, six months parallel group study. The flow chart of the study is reported in table 1. Participants initially will undergo 2 days of screening and testing. During the first visit patients will sign an informed consent, will undergo clinical assessment, pulmonary function testing, measurement of anthropometric data and body composition by bioimpedentiometry. They will perform a graded exercise test on a cycloergometer and will complete questionnaires to assess HRQoL (short form-36, SF-36) and functional abilities (health assessment questionnaire disability index, HAQ-DI). During the second visit, the participants will carry out the hand mobility in scleroderma test (HAMIS), six minutes walking test (6MWT), will undergo measurements of quadriceps and biceps strength, and handgrip test. After completion of testing and screening, patients who will meet the selection criteria will be randomly assigned to one of two groups 1) home-care rehabilitation group (HCRG); 2) control group (CG). The first group will begin a six months program of exercise training. The patients of the second group will be given generic recommendations to increase physical activity.

The patients in the first group, during a session in our outpatient clinic, will be instructed by a physiotherapist how to perform the physical exercise program at home. In particular, they will learn how to use the stationary bike and how to perform the exercises for upper limbs. Furthermore, the patient of the first group will be instructed how to fill in a card in which they will record the exercises performed daily. Throughout the first three months of the training period, the patients received a phone call from a physiotherapist once monthly, during which the adherence to exercise program will be reinforced. Particularly, it will be asked about the adherence to and the acceptance of exercise program, and the presence of side effects. Also, the control group will receive a phone call with the same schedule, but only in order to evaluate health status and to give a general recommendation about the positive effect of the aerobic exercise. From the third to the sixth month, both groups will not receive a monthly call, in order to evaluate the adherence to the program in the absence of supervision.

After 3 and 6 months, the subjects will undergo a complete 2 days of testing, using the same schedule described for a baseline.

The exercise program consists of aerobic exercise on a stationary bike, muscular endurance training of the upper limb and stretching exercises for finger joint motion. The exercise on the stationary bike and muscular endurance training will be performed on alternate days, three times a week.

A stationary cycle (Energetics ct220p, Neomark Sarl, Luxembourg) will be given to each patient for lower limb training. Each session will consist of three phases. In the first one, the patient will pedal for 5 minutes without inserting the brake. In the second phase, the patient will be instructed to set the brake at a load equal to 60% of the watts achieved at the peak of the maximal ergocycle exercise test. This phase consists in two periods of fifteen minutes divided by recovery interval of three minutes. It will be followed by five minutes of cool-down without load. The frequency of pedalling will be about 60 rotation/min during the second phase and less than 50 during the other phases.

For upper limbs training the patients will perform ten repetitions for three times that consists in lifting and lowering repeatedly a weight from the waist to the shoulders, alternating periods of exercise and three minutes of rest. The load will be calculated as the 60% of predicted 1-RM. Warm up and stretching of upper limbs, shoulders and neck will be performed before and after each exercise session respectively.

For the first two weeks, for both types of exercises of the program, the load will be reduced by 20%.

For finger stretching to the patients will be given written and illustrated instructions on self-administered exercises, and will be directed to perform it every day, both in the morning and in the evening.

During the rehabilitation period, the patients will report each day on a diary for each type of exercise whether the tasks were complete, partially or not executed which corresponds a score of 1, 0.5, 0 respectively.

The attendance rate at the training session will be calculated by the ratio between the amount of the score obtained from the diary and the scheduled sessions multiplied for 100.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of SSc according to the criteria of ACR
* no hospitalizations in the previous 3 months
* no change in anti-rheumatic treatment in the previous 3 months
* signed informed consent

Exclusion Criteria:

* heart failure staging in classes III or IV of New York Heart Association (NYHA)
* pulmonary hypertension, defined by echocardiogram as a right ventricular systolic pressure ≥ 45mmHg
* vital capacity (VC) ≤ 50% or diffusion lung capacity of carbon monoxide (DLCO) ≤ 30% of predicted values.
* renal failure defined as a calculated glomerular filtration rate (GFR) < 30ml/min, in agreement with the staging of International Federation of National Kidney Foundations
* inability to perform the rehabilitation program due to skeletal-muscle impairments or other illnesses
* pregnancy or planned pregnancy in the next 6 months
* psychiatric disorders that prevent collaboration and adherence at the rehabilitation the program, including drug abuse
* involvement in ongoing aerobic or anaerobic exercise programs

Drop out criteria:

* the demonstration of ischemic heart disease after cardiopulmonary exercise testing performed at baseline
* need to change the dosage or interruption of prostanoids used in the treatment of SSc during the 6 months of the treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Six minute walking test | Up to six months
  Evaluate aerobic capacity

SECONDARY OUTCOMES:
Maximum oxygen consumption (VO2max) | Up to six months
  Evaluate the maximum volume of oxygen that a human can consume in the unit of time, measured by cardiopulmonary test
Handgrip strength | Up to six months
  Handgrip strength will be measured in kilograms using a hydraulic hand-held dynamometer (Saehan Corp., Masan, Korea).Will be recorded, for each hand, the best result between three attempts.
Muscular strength of upper limbs | Up to six months
  Biceps strength will be measured in kilograms by an isometric forearm flexion using a dynamometer (Kern CH50K50, Kern&Sohn, Balingen, Germany) perpendicularly fixed on the floor. Will be recorded, for each arm, the best result between three attempts.
One repetition maximum (1-RM) of biceps strength | Up to six months
  One repetition maximum (1-RM) of biceps strength, expressed in kilograms, will be determinated by using the submaximal estimation method (predicted 1-RM) with the formula of Brzycke.
Muscular strength of lower limbs | Up to six months
  Quadriceps strength will be measured in kilograms by an isometric leg extension. The subject will be seated in an adjustable, straight-backed chair with the lower leg unsupported and the hip and knee flexed in a 90° angle, with an adjustable belt around the hips. Isometric leg extension strength will be measured by a dynamometer (Kern CH50K50, Kern & Sohn, Balingen, Germany) applied with a strap around the ankle just proximal to malleoli. Will be recorded, for each lower limb, the best result between three attempts.
Hand Mobility in Scleroderma test (HAMIS-test) | Up to six months
  Evaluate finger joint motion and hand function
Short Form - 36 (SF-36) | Up to six months
  It is a self-reported questionnaire for evaluating the health status. It contains 36 items, measuring quality of life with two summary measures, a physical component score (PCS) and a mental component score (MCS).
Health assessment questionnaire - disability index (HAQ-DI) | Up to six months
  This questionnaire indicates the extent of functional abilities. It consists in 20 items divided into eight categories. For each one of the items the score can range from 0 (lack of disability) to 3 (complete disability).
Adherence to exercise program, only for treatment group | Up to six months
  Evaluate the adherence, using a diary, during two periods of three months, one whit and one without supervision and reinforcement by phone call

CONTACTS AND LOCATIONS:
Overall Officials: Marcello Ferrari, Professor, Principal Investigator — Universita di Verona
Locations (1):
- Azienda Ospedaliera, SSO respiratory pathophysiology Unit, Verona, Verona, Italy/Verona, Italy

IPD SHARING:
Plan to Share IPD: Undecided